CLINICAL TRIAL: NCT05431959
Title: Evaluation of the Effect of Sulphur Mineral, Thermal Water on Skin Microbiome in Plaque Psoriasis, a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Tamás Bender, Professor of Medicine, Szeged University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZEGEDU
Record Dates: First submitted 2022-06-08; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Plaque Psoriasis
Keywords: balneotherapy; microbiome
MeSH Terms: interventions — Balneology

STUDY DESIGN:
Intervention Model Description: immersion in Lake Hévíz, 36℃ sulphur, carbonate, calcium, magnesium, hydrogen carbonate and very light radon-content thermal-mineral water 15 times in 3 weeks 30-minute therapy sessions. The total mineral substance of the water is 754 mg/l.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-controlled (Experimental): The skin microbiome was collected by swabbing method from the crook of the arm (normal skin) and the nearest plaque's surface.
  Balneotherapy in Lake Hévíz, 36℃ sulphur, carbonate, calcium, magnesium, hydrogen carbonate and very light radon-content thermal-mineral water 15 times in 3 weeks 30-minute therapy sessions. The total mineral substance of the water is 754 mg/l.
  Interventions: Other: balneotherapy

INTERVENTIONS:
Other: balneotherapy — immersion in Lake Hévíz, 36℃ sulphur, carbonate, calcium, magnesium, hydrogen carbonate and very light radon-content thermal-mineral water 15 times in 3 weeks 30-minute therapy sessions. The total mineral substance of the water is 754 mg/l.

SUMMARY:
In this study the effects of balneotherapy in Lake Hévíz, 36℃ sulphur, carbonate, calcium, magnesium, hydrogen carbonate and very light radon-content thermal, mineral water on skin microbiome and Psoriasis Area and Severity Index (PASI) in patients with plaque psoriasis

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory skin disease. It is associated with several important medical conditions, including psoriatic arthritis, and cardiometabolic syndrome. Its most common form, chronic plaque.The aim of this study is to evaluate how Lake Hévíz sulphur thermal mineral water therapy influences the composition of microbial communities that colonizes skin in patients with psoriasis, and the extent and severity of skin symptoms of psoriasis.

The planned participants number is 16 outpatients between 18 and 70 years of age with mild to moderate psoriasis. The balneotherapy takes place in Lake Hévíz, five times a week for three weeks.

The skin microbiome is collected from two different place by swabbing method from the patient. One sample is collected from the normal skin, which is not affected by psoriasis (crook of the arm), the second sample is collected from psoriatic plaque of the elbow. The samples is processed for a sequence-based microbiome analysis.

The skin microbiome is evaluated by the analysis of the sample metagenome compositions, and the activity of psoriasis is evaluated on The Psoriasis Area and Severity Index (PASI), is taken at week 0., at week 3.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque psoriasis for at least 6 months before the Baseline Visit
* Subject has stable mild to moderate plaque psoriasis

Exclusion Criteria:

* subject has systemic therapy for plaque psoriasis
* balneotherapy within 3 months prior the enrollement
* systemic/local glucocorticoid therapy within 1 month prior the enrollment
* general contraindications to balneotherapy: decompensated cardiovasculardisease; unstable hypertension, angina pectoris; uncontrolled endocrinedisease (hyperthyroidism, hyperparathyroidism); other uncontrolledand unstable metabolic disorders (diabetes mellitus, hyperuricaemia,hyperlipoproteinaemia); acute febrile infections; cutaneous suppuration;pregnancy; decompensated psychosis/neurosis, malignancy, urine and stool incontinent, unconsciousness, alcoholic influence, and lack of compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-07-25 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
1. Alpha diversity | baseline to week 3
  Determination of microbiom in samples (bacterial DNA are isolated from the skin to determine the microbial composition) Number of species with Shannon-, Simpson and Chao1 indexes
2. Change in microbiota diversity before and after balneotherapy treatment | baseline to week 3
  Change in alpha diversity before and after treatment:to compare normal samples before and after treatment, to compare psoriasis samples before and after treatment and the comparison of normal and psoriasis samples before treatment.Differences in genus abundances to determine with the core function of the microbiome R package (Lahti et al., 2019), with detection 100 and prevalence 0.1.

SECONDARY OUTCOMES:
1. Beta diversity | baseline to week 3
  Inter-sample genus composition differences by the Bray-Curtis beta-diversity metric
2. The Psoriasis Area and Severity Index (PASI) allows evaluating the extent and severity of skin symptoms of psoriasis. | baseline to week 3
  Percentage of Participants With a 50% Reduction From Baseline Psoriasis Area and Severity Index (PASI 50) at Week 3. The PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 50 is defined as at least a 50% reduction in PASI score compared with the Baseline PASI score.

CONTACTS AND LOCATIONS:
Locations (2):
- Hungary (2):
  - Tamas Bender, Budapest
  - Ágota Kulisch, MD, PhD, Hévíz

IPD SHARING:
Plan to Share IPD: No
In this study the effects of balneotherapy in Lake Hévíz, 36℃ sulphur, carbonate, calcium, magnesium, hydrogen carbonate and very light radon-content thermal, mineral water on skin microbiome and Psoriasis Area and Severity Index (PASI) in patients with plaque psoriasis.

REFERENCES:
- [Background] De Pessemier B, Grine L, Debaere M, Maes A, Paetzold B, Callewaert C. Gut-Skin Axis: Current Knowledge of the Interrelationship between Microbial Dysbiosis and Skin Conditions. Microorganisms. 2021 Feb 11;9(2):353. doi: 10.3390/microorganisms9020353. PMID 33670115
- [Background] Martin R, Henley JB, Sarrazin P, Seite S. Skin Microbiome in Patients With Psoriasis Before and After Balneotherapy at the Thermal Care Center of La Roche-Posay. J Drugs Dermatol. 2015 Dec;14(12):1400-5. PMID 26659932
- [Background] Peinemann F, Harari M, Peternel S, Chan T, Chan D, Labeit AM, Gambichler T. Indoor balneophototherapy for chronic plaque psoriasis: Abridged Cochrane Review. Dermatol Ther. 2021 Jan;34(1):e14588. doi: 10.1111/dth.14588. Epub 2020 Dec 2. PMID 33236826
- [Result] Griffiths CEM, Armstrong AW, Gudjonsson JE, Barker JNWN. Psoriasis. Lancet. 2021 Apr 3;397(10281):1301-1315. doi: 10.1016/S0140-6736(20)32549-6. PMID 33812489
- [Result] Darlenski R, Bogdanov I, Kacheva M, Zheleva D, Demerdjieva Z, Hristakieva E, Fluhr JW, Tsankov N. Disease severity, patient-reported outcomes and skin hydration improve during balneotherapy with hydrocarbonate- and sulphur-rich water of psoriasis. J Eur Acad Dermatol Venereol. 2021 Mar;35(3):e196-e198. doi: 10.1111/jdv.16908. Epub 2020 Sep 17. No abstract available. PMID 32869298